CLINICAL TRIAL: NCT00773578
Title: Impact of Environmental Tobacco Smoke on Exhaled Nitric Oxide and on Biomarkers of Nasal Inflammation in Atopic Asthmatic Children
Brief Title: Exhaled Nitric Oxide and Nasal Lavage Fluid
Acronym: NOLN
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Yannick Vacher, Department Clinical Research of Developpement
Other Study IDs: P070201; AOR05005
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Asthma
Keywords: Children; Tobacco smoke exposure; Exhaled nitric oxide; Nasal lavage; Cytokines
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: atopic asthmatic children exposed to environmental tobacco smoke
  Interventions: Device: Measurement of exhaled nitric oxide (eNO); Device: Measurement of biomarkers of nasal inflammation
- 2: atopic asthmatic children unexposed to environmental tobacco smoke
  Interventions: Device: Measurement of exhaled nitric oxide (eNO); Device: Measurement of biomarkers of nasal inflammation

INTERVENTIONS:
Device: Measurement of exhaled nitric oxide (eNO) — Chemiluminescence NO analyzer Measurement of lung function (spirometry)
Device: Measurement of biomarkers of nasal inflammation — Nasal lavage

SUMMARY:
The allergic respiratory diseases such as asthma or allergic rhinitis are the main chronic diseases in children. The airway inflammation plays an important role in their pathophysiology. Several epidemiological studies show that environmental tobacco smoke (ETS) exacerbates the symptoms of asthma and allergies.

The aim of this study is to assess the impact of environmental tobacco smoke on the measurement of exhaled nitric oxide (eNO) and biomarkers of nasal inflammation in atopic asthmatic children.

DETAILED DESCRIPTION:
Type of study :

This study is a epidemiological observation study type exposed or unexposed to environmental tobacco smoke.

Methods :

The eNO is determined by a method On-line, at a rate expiratory 50 mL / s, using a chemiluminescence NO analyzer, before the allergy assessment (skin tests and assay of serum total and specific IgE ) and measurement of lung function (spirometry). Nasal lavage is performed by using a validated technique . Cells are counted and differentiated after Giemsa staining. We measured 1-anti-trypsin, neutrophil elastase, albumin, urea, IL4 , IL6, IL8 and IL13. Exposure to ETS is assessed by questionnaire to the parents. Statistical analysis include a narrative strand to verify the normality of distribution and an analytical analysis, including a bivariate followed by a multivariate analysis by multiple linear regression and / or logistic regression to model concentrations of biomarkers of inflammation and adjustment variables such as age, sex, atopic status, eosinophilia and severity of asthma.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 5 years
* Atopic, persistent mild and moderate Asthmatic Children (GINA 2 and 3)

Exclusion Criteria:

* Child with asthma medication asthma used in the previous 15 days (oral or inhaled corticosteroids, leukotriene antagonist)
* Recent asthma attack (day of hospitalization or 15 days earlier)
* Upper respiratory infection (4 weeks) and low (2 weeks)
* Active smoking (teenager)

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Atopic asthmatic children followed in the Asthma Center, Trousseau Hospital, Paris
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Assessment of the impact of environmental tobacco smoke on the measurement of exhaled nitric oxide and the nasal inflammation biomarkers, in atopic asthmatic children aged over 5 years | at the inclusion visit

SECONDARY OUTCOMES:
Evaluation of the possible association between nasal inflammation (objectified by the determination of biomarkers in the nasal lavage fluid) and bronchial (measurement of exhaled nitric oxide). | At the inclusion visit

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyne JUST, MdPh, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Trousseau, Paris, France